CLINICAL TRIAL: NCT06897215
Title: A Sequential Cohort Study Exploring Gelclair in the Management of Oral Mucostitis (OM) in Patients Receiving Radical Radiation for Head and Neck Cancer (GOMS)
Brief Title: A Sequential Cohort Study Exploring GELCLAIR in the Management of Oral Mucositis in Patients Receiving Radical Radiation for Head and Neck Cancer
Acronym: GOMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Murali Rajaraman, Radiation Oncologist, Nova Scotia Health Authority
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 71716
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Oral Mucositis Due to Radiation
Keywords: Oral Mucositis; Radiation toxicity; Gelclair; hyaluronic acid hydrogel
MeSH Terms: conditions — Stomatitis; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: The first cohort of patients (16) will be evaluated for oral mucositis (OM) development and management while undergoing current standard of care which includes lidocaine-based mouthwashes as initial treatment. The subsequent (experimental) cohort of patients (32) will begin treatment with Gelclair once significant OM develops with the same evaluation parameters as the previous (control) cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (No Intervention): The first cohort of patients (16) will be evaluated for oral mucositis (OM) development and management while undergoing current standard of care which includes lidocaine-based mouthwashes as initial treatment and weekly assessments during 6-7 weeks of radiation treatment up to and including 4 weeks post-radiation treatment.
- Experimental Cohort (Experimental): The subsequent (experimental) cohort of patients (32) will begin treatment with Gelclair once significant OM develops with the same evaluation parameters as the previous (control) cohort. Gelclair be used at the onset of Grade 2 OM topically to be swished in the oral cavity and then spit 3 times a daily during treatment and until OM symptoms resolve which is usually at least 4 weeks after completion of RT.
  Interventions: Device: Hyaluronic acid hydrogel

INTERVENTIONS:
Device: Hyaluronic acid hydrogel — Assigned to the Experimental Cohort once OM grade 2.0 presents, Gelclair is a hyaluronic acid hydrogel that acts as a protective film in the management of OM. This product is used internationally and has been recently approved by Health Canada as a Class 2 Medical Device with an indication to manage the symptoms of OM caused by radiotherapy and chemotherapy.
  Other Names: Gelclair
  Arms: Experimental Cohort

SUMMARY:
The goal of this clinical trial is to learn if Gelclair lubricant gel can help manage Oral Mucositis (OM) among Oropharyngeal and Oral cavity cancer patients receiving radiation treatment. The main questions it aims to answer are:

1. Does Gelclair help to manage the symptoms of OM and decrease its severity?
2. What do participants report as the maximum levels of pain and difficulties with swallowing?

Researchers will compare Gelclair to the standard of care mouthwash treatment for OM (currently used for all patients with symptomatic OM) to see if Gelclair is helpful in managing oral mucositis.

For the cohort using Gelclair, participants will:

1. Take the prescribed treatment for OM (Gelclair or Oncology mouthwash) once it is diagnosed, up to and including 4 weeks after radiation completes.
2. Complete a weekly survey about their OM symptoms up to and including 4 weeks after radiation completes.

2. Report any problems experienced with prescribed treatment for OM (Gelclair or mouthwash).

The same data will be collected for the cohort using standard of care mouthwash for comparison.

DETAILED DESCRIPTION:
Radiotherapy (RT) induced mucositis, including oral mucositis (OM), is the most common high-grade toxicity observed during high dose RT for Head and Neck Cancer (HNC). Prevention usually consists of adhering to oral care protocols, avoiding irritants, and avoiding mucosal hot spots in the RT plan. Once it occurs, analgesic treatments include various mixtures of pain relief mouthwashes, NSAIDS, opioids, and steroids and antifungals as indicated.

Mucoadhesive topical coating agents have been used to treat RT induced OM.

Study eligible patients will be offered participation after clinic consultation has taken place. They will be detailed provided study information and if they consent in writing, will be assigned to the standard of care cohort (16 patients) and the experimental cohort (32 patients) in a sequential format.

The first cohort of 16 patients will be evaluated for oral mucositis (OM) using CTCAE V5 criteria and Patient Reported Outcome questionnaires while undergoing management with current standard of care for symptomatic OM which includes lidocaine-based mouthwashes as initial treatment. The subsequent (experimental) cohort of 32 patients will begin treatment with Gelclair once symptomatic OM develops with the same evaluation parameters as the previous (control) cohort. Gelclair is a hyaluronic acid hydrogel that acts as a protective film in the management of OM. This product is used internationally and has been recently approved by Health Canada as a Class 2 Medical Device with an indication to manage the symptoms of OM caused by radiotherapy and chemotherapy.

After collection of baseline data (including age, sex, cancer diagnosis and staging, relevant past medical history, treatment plan, weight, nutrional status), weekly data (includes OM grading, Patient Reported Outcome for OM, weight, analgesic requirements, parenteral nutrional requirements, side effects, adherence to protocol) during radiation therapy (RT) and for 4 weeks after RT completion is recorded.

Upon study completion, analysis will be aimed at the following outcomes:

Primary Objective: Explore the effectiveness of GelClair versus SOC mouth wash in the management of symptomatic radiation-induced OM.

Secondary Objectives: Patient reported outcomes (PRO) for maximum levels reached of odynophagia and dysphagia (assessed weekly from RT start until 4 weeks after completion)

Other measurement outcomes include time to initiation of opioid (or increase in baseline dose) measured in days, weight loss, treatment delays / modifications due to OM, requirement for feeding tube, adherence to treatment protocol, cost analysis for SOC mouthwash versus GelClair based on total days use of each agent.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary mucosal squamous cell carcinoma of the oropharynx or oral cavity
* Treatment plan includes at least 60Gy of daily radiotherapy, with or without concurrent chemotherapy
* Highly likely to develop OM CTCAE v5.0, grade 2
* Can read and understand English

Exclusion Criteria:

- Patients who already have parenteral feeding tubes prescribed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the effectiveness of GelClair versus SOC mouth wash in the management of symptomatic OM. | From enrollment up to and including 4 weeks after treatment completion.
  The reduction of maximum Grade 2 (CTCAE V5.0) oral mucositis will be compared between the two cohorts.

SECONDARY OUTCOMES:
Time to Initiation of Opioid or Increase in baseline dose | From enrollment up to and including 4 weeks after radiation treatment completes.
  Quantitative comparison between cohorts calculating (in days) the need to increase or change participant's management of OM.
Changes in Weight | From enrollment up to and including 4 weeks after radiation treatment completes.
  Quantitative comparison between cohorts calculating change in weight weight (in kgs) in participants.
Significant treatment delays/modifications | From enrollment up to and including 4 weeks after radiation treatment completes.
  Measured as a yes/no flag comparing totals across the cohorts
Requirement for feeding tube | From enrollment up to and including 4 weeks after radiation treatment completes.
  Quantitative comparison between cohorts of total number of patients requiring a new feeding tube during the course of radiation treatment.
Rate of adherence to treatment protocol using Patient Reported Outcomes | From enrollment up to and including 4 weeks after radiation treatment completes.
  Quantitative comparison between cohorts for compliance with prescribed treatment of OM measured weekly.

CONTACTS AND LOCATIONS:
Overall Officials: Murali Rajaraman, Principal Investigator — Nova Scotia Health; Derek Wilke, Principal Investigator — Nova Scotia Health

IPD SHARING:
Plan to Share IPD: No
This is a single center study and IPD will not be shared with anyone outside the study personnel at this center.